CLINICAL TRIAL: NCT02840721
Title: A PHASE 2A, MULTICENTER, SINGLE ARM, OPEN- LABEL, TWO-STAGE, STUDY TO EVALUATE THE EFFICACY, SAFETY, TOLERABILITY AND PHARMACOKINETICS OF PF-06480605 IN SUBJECTS WITH MODERATE TO SEVERE ULCERATIVE COLITIS
Brief Title: Safety, Efficacy, and Tolerability Study of PF-06480605 in Subjects With Moderate to Severe Ulcerative Colitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Telavant, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7541002; TUSCANY (Other: Alias Study Number); 2016-001158-16 (EudraCT Number)
Record Dates: First submitted 2016-06-27; First posted 2016-07-21 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06480605 (Experimental): PF-06480605 500 mg IV Q2W X 7 doses
  Interventions: Drug: PF-06480605

INTERVENTIONS:
Drug: PF-06480605 — PF-06480605 500 mg IV Q2W x 7 Doses

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of PF-06480605 in subjects with moderate to severe ulcerative colitis.

DETAILED DESCRIPTION:
This is a Phase 2a, single arm, two-stage study in subjects with moderate to severe ulcerative colitis. Subjects will receive 500 mg of PF-06480605 intravenously every 2 weeks for a total of 7 doses. Blood, stool, and tissue samples will be collected at various time points throughout the study to evaluate safety, tolerability, efficacy, pharmacokinetics, and immunogenicity. Duration of participation for subjects will be approximately 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between ≥ 18 and ≤ 75 years of age at the time of informed consent
* Male subjects able to father children and female subjects of childbearing potential must agree to use two highly effective methods of contraception throughout the study and until the Week 26 visit
* Diagnosis of ulcerative colitis for ≥ 4 months
* Subjects with moderate to severe active ulcerative colitis as defined by screening colonoscopy with total Mayo score of ≥ 6, with rectal bleeding subscore of ≥ 1, and an endoscopic subscore of ≥ 2 on the Mayo
* Active disease beyond the rectum (> 15 cm of active disease at the screening colonoscopy)
* Must have inadequate response to, loss of response to, or intolerance to at least one conventional therapy for ulcerative colitis such as: Steroids; Immunosuppressants (AZA, 6-MP, or MTX); Anti -TNF inhibitors (eg, infliximab, adalimumab, or golimumab); Anti-integrin inhibitors (eg, vedolizumab).
* Subjects currently receiving the following treatment are eligible provided they have been on stable doses of Oral 5-ASA or sulfasalazine for at least 4 weeks prior to baseline; oral corticosteroids stable dose for at least 2 weeks prior to baseline; 6-MP or AZA stable dose for 8 weeks prior to baseline.

Exclusion Criteria:

* Diagnosis of indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis, microscopic colitis or Crohn's Disease. Subjects with clinical findings suggestive of Crohn's disease (eg, fistulae, granulomas on biopsy) are also excluded.
* Subjects with colonic dysplasia or neoplasia, toxic megacolon, primary sclerosing cholangitis, known colonic stricture, history of colonic or small bowel stoma, history of colonic or small bowel obstruction or resection
* Presence of active enteric infections (positive stool culture and sensitivity)
* Known history of HIV based on documented history with positive serological test, or positive HIV serologic test at screening
* Presence of a transplanted organ
* Cancer or history of cancer or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell or squamous cell carcinoma that has been treated with no evidence of recurrence);
* Acute coronary syndrome (eg., myocardial infarction, unstable angina pectoris);
* Any history of cerebrovascular disease within 24 weeks before screening;
* Subject with current or a history of QT prolongation
* Class III or Class IV heart failure
* Prior evidence of liver injury or toxicity due to methotrexate
* Abnormality in hematology and/or chemistry profiles during screening (as detailed in the protocol)
* Subjects receiving the following therapies within the designated time period:

  * > 9 mg/day of oral budesonide or >20 mg/day prednisone or equivalent within 2 weeks prior to baseline
  * IV, IM (parenteral), or topical (rectal) treatment of 5-ASA or corticosteroid enemas/suppositories within 2 weeks prior to baseline
  * Biologics including anti-TNF inhibitors as described: Infliximab, Adalimumab, or Golimumab within 8 weeks prior to baseline
  * Anti-integrin inhibitors (eg, vedolizumab) within 12 weeks prior to baseline
  * Other investigational procedures or products, or live attenuated vaccine within 30 days prior to baseline.
* Current or history (within 2 years) of serious psychiatric disease or alcohol or drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (12):
  - Surgery Center of Aventura, Aventura, Florida
  - Venture Ambulatory Surgical Center, North Miami Beach, Florida
  - FQL Research, LLC, Pembroke Pines, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - NYU Langone Nassau Gastroenterology Associates, Great Neck, New York
  - New York Presbyterian Hospital-Weill Cornell Medical College, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Weill Cornell Medicine, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Allegiance Research Specialists, LLC, Wauwatosa, Wisconsin
- Belgium (3):
  - UZ Leuven (University Hospital Leuven) - Pharmacy Clinical Trials, Leuven
  - UZ Leuven (University Hospital Leuven) - Radiology Department, Leuven
  - UZ Leuven (University Hospital Leuven), Campus Gasthuisberg, Leuven
- Italy (3):
  - AOU Mater Domini - Univ."Magna Graecia" di Catanzaro - Campus Venuta - U.O Fisiopatologia Digestiva, Catanzaro, CZ
  - ISTITUTO CLINICO HUMANITAS Sezione Autonoma di Malattie Infiammatorie Croniche Intestinali, Rozzano, Milan (MI)
  - Policlinico Universitario Campus Biomedico, Roma, RM
- Netherlands (3):
  - Academic Medical Center, Apotheek-Kenniscentrum Geneesmiddelenonderzoek, Amsterdam, North Holland
  - Academic Medical Centre, Department of Radiology, Amsterdam, North Holland
  - Academic Medical Centre, Dept. of Gastroenterology, Amsterdam, North Holland
- Poland (5):
  - SPZOZ WSzZ im. Jedrzeja. Sniadeckiego W Bialymstoku Oddzial Chorob Wewnetrznych i Gastroenterologii, Bialystok
  - Centrum Endoskopii Zabiegowej, Poradnia Chorob Jelitowych Szpital Uniwersytecki nr 2 im Jana Biziela, Bydgoszcz
  - Piotr Walczak Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - SANTA FAMILIA Centrum Badan Profilaktyki i Leczenia, Lodz
  - Endoskopia Sp. z.o.o., Sopot
- South Korea (2):
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Danese S, Klopocka M, Scherl EJ, Romatowski J, Allegretti JR, Peeva E, Vincent MS, Schoenbeck U, Ye Z, Hassan-Zahraee M, Rath N, Li G, Neelakantan S, Banfield C, Lepsy C, Chandra DE, Hung KE. Anti-TL1A Antibody PF-06480605 Safety and Efficacy for Ulcerative Colitis: A Phase 2a Single-Arm Study. Clin Gastroenterol Hepatol. 2021 Nov;19(11):2324-2332.e6. doi: 10.1016/j.cgh.2021.06.011. Epub 2021 Jun 12. PMID 34126262
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7541002

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-06480605 500 mg IV: Participants received PF-06480605 500 mg intravenously once every 2 weeks (Q2W) for a total of 7 doses (i.e., 12-week treatment period), and then were followed up for additional 14 weeks after the last dose of PF-06480605.
Period: Treatment Period
Arm/Group | PF-06480605 500 mg IV
Started | 50
Completed | 49
Not Completed | 1
Not completed — Adverse Event | 1
Period: Follow-Up
Arm/Group | PF-06480605 500 mg IV
Started | 49
Completed | 42
Not Completed | 7
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 4
Not completed — Withdrawal of Consent | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled in the study.
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (14.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48
  Asian | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events, Serious Adverse Events, and Who Withdrew Due to Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. A serious AE (SAE) was any untoward medical occurrence at any dose that (1) resulted in death; (2) was life-threatening (immediate risk of death); (3) required inpatient hospitalization or prolongation of existing hospitalization; (4) resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); (5) resulted in congenital anomaly/birth defect. A treatment-emergent AE (TEAE) was defined as an event that emerged during treatment having been absent pre-treatment, or worsened relative to the pre-treatment state. Causality to study treatment was determined by the investigator.
Time Frame: Day 1 up to final onsite visit (Week 26)
Population: The analysis population included all participants who received at least 1 dose of PF-06480605.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 50
Participants
  All-causality AEs | 33
  All-causality SAEs | 3
  Treatment-related AEs | 8
  Treatment-related SAEs | 1
  Withdrew due to AEs | 1

2. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: The following parameters were evaluated: hematology (hemoglobin, hematocrit, erythrocytes, erythrocyte mean corpuscular volume, platelets, leukocytes, lymphocytes, neutrophils, basophils, eosinophils, monocytes, activated partial thromboplastin time, and prothrombin time), clinical chemistry (bilirubin, direct bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, protein, albumin, blood urea nitrogen, creatinine, urate, sodium, potassium, chloride, calcium, glucose, and creatine kinase), and urinalysis (urine glucose, ketones, urine protein, urine hemoglobin, nitrite, leukocyte esterase, urine erythrocytes, urine leukocytes, hyaline casts, and bacteria).
Time Frame: Day 1 up to final onsite visit (Week 26)
Population: The analysis population included all participants who received at least 1 dose of PF-06480605.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 50
Participants | 38

3. Primary Outcome: Number of Participants With Vital Signs Data Meeting Pre-specified Criteria
Description: Vital signs evaluation included sitting diastolic blood pressure (DBP), systolic blood pressure (SBP), and pulse rate. Sitting blood pressure was measured with the participant's arm supported at the level of the heart, and recorded to the nearest millimeters of mercury (mm Hg). The same size BP cuff which had been properly sized and calibrated was used to measure BP each time. Number of participants with vital signs data meeting pre-specified criteria is presented.
Time Frame: Baseline up to final onsite visit (Week 26)
Population: The analysis population included all participants who received at least 1 dose of PF-06480605.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 50
Participants
  Sitting DBP <50 mm Hg | 1
  Sitting SBP <90 mm Hg | 4
  Sitting pulse rate <40 beats per minute (bpm) | 0
  Sitting pulse rate >120 bpm | 1
  Sitting DBP increase from baseline >=20 mm Hg | 2
  Sitting SBP increase from baseline >=30 mm Hg | 5
  Sitting DBP decrease from baseline >=20 mm Hg | 7
  Sitting SBP decrease from baseline >=30 mm Hg | 1

4. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-specified Criteria
Description: All scheduled 12-lead ECGs were performed after the participant had rested quietly for at least 10 minutes in a supine position. Number of participants with ECG data meeting pre-specified criteria is presented.
Time Frame: Baseline up to final onsite visit (Week 26)
Population: The analysis population included all participants who received at least 1 dose of PF-06480605 and had both baseline and at least 1 post-baseline ECG evaluation performed.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 49
Participants
  PR interval >=300 milliseconds (msec) | 0
  QRS duration >=140 msec | 0
  QT interval >=500 msec | 0
  QTcF interval: 450 to <480 msec | 5
  QTcF interval: 480 to <500 msec | 0
  QTcF interval: >=500 msec | 0
  PR interval increase from baseline >=25%/50% | 0
  QRS duration increase from baseline >=50% | 0
  QTcF increase from baseline: 30 to <60 msec | 9
  QTcF increase from baseline: >=60 msec | 1

5. Primary Outcome: Percentage of Participants Achieving Endoscopic Improvement at Week 14, Based on Uniformly Minimum-Variance Unbiased Estimator (UMVUE) - Per Protocol Analysis Set
Description: Endoscopic improvement at Week 14 was defined as Mayo endoscopic sub-score of 0 or 1, and without friability. The Mayo scoring system was used to assess ulcerative colitis activity, and it ranges from 0 to 12, calculated as sum of 4 sub-scores, with higher scores indicating more severe disease. The 4 sub-scores are stool frequency (0=normal number of stools; 1=1 to 2 stools more than normal; 2=3 to 4 stools more than normal; 3= 5 or more stools more than normal); rectal bleeding (0=no blood seen; 1=streaks of blood with stools less than half the time; 2=obvious blood with stool most of the time; 3=blood alone passes); findings on endoscopy (0=normal or inactive disease; 1=mild disease [erythema, decreased vascular pattern, mild friability]; 2=moderate disease [marked erythema, lack of vascular pattern, friability, erosions]; 3=severe disease [spontaneous bleeding, ulceration]); and physician's global assessment (0=normal; 1=mild disease; 2=moderate disease; 3=severe disease).
Time Frame: Week 14
Population: The analysis population included all participants who were eligible for enrollment, not a major protocol violator, with at least 6 out of 7 planned doses received and a final colonoscopy at Week 14.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 45
percentage of participants | 38.20 [23.82 to 53.68]

6. Secondary Outcome: Percentage of Participants Achieving Remission at Week 14 - Full Analysis Set
Description: Remission: total Mayo score <=2 with no individual subscore >1. Mayo scoring system was used to assess ulcerative colitis activity (range: 0 to 12, calculated as sum of 4 subscores, higher scores indicating more severe disease). The 4 subscores are stool frequency (0=normal number of stools; 1=1 to 2 stools more than normal; 2= 3 to 4 stools more than normal; 3= 5 or more stools more than normal); rectal bleeding (0=no blood seen; 1=streaks of blood with stools less than half the time; 2=obvious blood with stool most of the time; 3=blood alone passes); findings on modified endoscopy (0=normal or inactive disease; 1=mild disease [erythema, decreased vascular pattern, no friability]; 2=moderate disease [marked erythema, lack of vascular pattern, friability, erosions]; 3=severe disease [spontaneous bleeding, ulceration]); and physician's global assessment (0=normal; 1=mild disease; 2=moderate disease; 3=severe disease).
Time Frame: Week 14
Population: The analysis population included all participants who received at least 1 dose of PF-06480605.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 50
percentage of participants | 24.00 [13.06 to 38.17]

7. Secondary Outcome: Percentage of Participants Achieving Remission at Week 14 - Per Protocol Analysis Set
Description: as for outcome 6
Time Frame: Week 14
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 45
percentage of participants | 26.67 [14.60 to 41.94]

8. Secondary Outcome: Percentage of Participants Achieving Endoscopic Remission at Week 14 - Full Analysis Set
Description: Endoscopic remission at Week 14 was defined as Mayo endoscopic sub-score of 0. The Mayo scoring system was used to assess ulcerative colitis activity, and it ranges from 0 to 12, calculated as sum of 4 sub-scores, with higher scores indicating more severe disease. The 4 sub-scores are stool frequency (0=normal number of stools; 1=1 to 2 stools more than normal; 2= 3 to 4 stools more than normal; 3= 5 or more stools more than normal); rectal bleeding (0=no blood seen; 1=streaks of blood with stools less than half the time; 2=obvious blood with stool most of the time; 3=blood alone passes); findings on endoscopy (0=normal or inactive disease; 1=mild disease [erythema, decreased vascular pattern, mild friability]; 2=moderate disease [marked erythema, lack of vascular pattern, friability, erosions]; 3=severe disease [spontaneous bleeding, ulceration]); and physician's global assessment (0=normal; 1=mild disease; 2=moderate disease; 3=severe disease).
Time Frame: Week 14
Population: The analysis population included all participants who received at least 1 dose of PF-06480605.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 50
percentage of participants | 10.00 [3.33 to 21.81]

9. Secondary Outcome: Maximum Serum Concentration (Cmax) of PF-06480605
Description: Maximum serum concentration (Cmax) of PF-06480605 was observed directly from data.
Time Frame: 30 minutes pre-dose and 1 hour post-dose on Day 85
Population: The analysis population included all enrolled participants who received at least 1 dose of PF-06480605 and in whom at least 1 concentration value was reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms (ng)/milliliters (mL)
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 44
nanograms (ng)/milliliters (mL) | 263400 (54)

10. Secondary Outcome: Average Serum Concentration (Cav) of PF-06480605
Description: Average serum concentration (Cav) of PF-06480605 was calculated as AUCtau/tau, where tau was the dosing interval (tau=14 days), and AUCtau was the area under the concentration-time profile from time 0 to time tau.
Time Frame: 30 minutes pre-dose and 1 hour post-dose on Day 85
Population: The analysis population included all enrolled participants who received at least 1 dose of PF-06480605 and had at least 1 derived value of a specific pharmacokinetic (PK) parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms (ng)/milliliters (mL)
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 44
nanograms (ng)/milliliters (mL) | 171400 (45)

11. Secondary Outcome: Lowest Serum Concentration (Cmin) of PF-06480605
Description: Lowest serum concentration (Cmin) of PF-06480605 was observed directly from data.
Time Frame: 30 minutes pre-dose and 1 hour post-dose on Day 85
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 44
ng/mL | 87650 (50)

12. Secondary Outcome: Area Under the Concentration-time Profile From Time Zero to Time Tau (AUCtau) of PF-06480605
Description: AUCtau of PF-06480605 was calculated using linear/log trapezoidal method; tau was the dosing interval (=14 days).
Time Frame: 30 minutes pre-dose and 1 hour post-dose on Day 85
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 44
ng.hr/mL | 57610000 (45)

13. Secondary Outcome: Percentage of Participants Who Developed Anti-drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs)
Description: Serum samples were analyzed using a new ADA assay with acid pre-treatment followed by a more drug-tolerant cell-based NAb assay. For ADA assay with acid pre-treatment, the sample was deemed positive if log titer >=1.30; for cell-based NAb assay, the sample was deemed positive if log titer >=0.699.
Time Frame: Day 1 up to final onsite visit (Week 26)
Population: The analysis population included all enrolled participants who received at least 1 dose of PF 06480605 with at least 1 post-treatment ADA determination.
Measure: Number; unit: percentage of participants
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 50
percentage of participants
  ADA | 82.0
  NAb | 10.0

14. Secondary Outcome: Change From Baseline in Fecal Calprotectin
Description: Fecal calprotectin has been used to detect intestinal inflammation (colitis or enteritis) and can serve as a biomarker for inflammatory bowel diseases. Elevated fecal calprotectin levels indicate migration of neutrophils into the intestinal mucosa, which occurs during intestinal inflammation.
Time Frame: Baseline, Weeks 2, 8, 12 and 26
Population: The analysis population included all participants who received at least 1 dose of PF 06480605 with at least 1 fecal calprotectin measurement.
Measure: Mean (Standard Deviation); unit: micrograms/grams
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 48
micrograms/grams
  Baseline | 3662.25 (3556.331)
  Week 2 change from baseline: number analyzed (Participants) | 46
  Week 2 change from baseline | -1861.38 (3565.861)
  Week 8 change from baseline: number analyzed (Participants) | 45
  Week 8 change from baseline | -2509.43 (3751.843)
  Week 12 change from baseline: number analyzed (Participants) | 42
  Week 12 change from baseline | -2844.26 (3623.922)
  Week 26 change from baseline: number analyzed (Participants) | 42
  Week 26 change from baseline | -2726.97 (3673.063)

15. Secondary Outcome: Change From Baseline in High Sensitivity C-reactive Protein (HsCRP)
Description: HsCRP is used mainly as a marker of inflammation.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, and 26
Population: The analysis population included all participants who received at least 1 dose of PF 06480605 with 1 hsCRP measurement.
Measure: Mean (Standard Deviation); unit: micrograms/deciliter
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 48
micrograms/deciliter
  Baseline | 0.9316 (1.15545)
  Week 2 change from baseline: number analyzed (Participants) | 46
  Week 2 change from baseline | -0.2136 (1.43785)
  Week 4 change from baseline: number analyzed (Participants) | 45
  Week 4 change from baseline | -0.4883 (1.10820)
  Week 6 change from baseline: number analyzed (Participants) | 47
  Week 6 change from baseline | -0.3314 (1.39605)
  Week 8 change from baseline: number analyzed (Participants) | 47
  Week 8 change from baseline | -0.4875 (1.00870)
  Week 10 change from baseline: number analyzed (Participants) | 45
  Week 10 change from baseline | -0.5738 (0.97608)
  Week 12 change from baseline: number analyzed (Participants) | 42
  Week 12 change from baseline | -0.4242 (1.18416)
  Week 14 change from baseline: number analyzed (Participants) | 42
  Week 14 change from baseline | -0.3983 (1.21181)
  Week 16 change from baseline: number analyzed (Participants) | 42
  Week 16 change from baseline | -0.5070 (1.37798)
  Week 20 change from baseline: number analyzed (Participants) | 42
  Week 20 change from baseline | -0.4728 (1.11950)
  Week 24 change from baseline: number analyzed (Participants) | 39
  Week 24 change from baseline | -0.5334 (1.03224)
  Week 26 change from baseline: number analyzed (Participants) | 40
  Week 26 change from baseline | -0.3453 (1.37576)

16. Secondary Outcome: Change From Baseline in Serum Total Soluable Tumor Necrosis Factor-like Ligand 1A (sTL1A)
Description: TL1A is a member of the tumor necrosis factor (TNF) family of cytokines. The investigational product of this study PF-06480605 is a fully human neutralizing antibody against TL1A.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, and 26
Population: The analysis population included all participants who received at least 1 dose of PF 06480605 with 1 sTL1A measurement.
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | PF-06480605 500 mg IV
Number analyzed (Participants) | 50
picograms/mL
  Baseline: number analyzed (Participants) | 47
  Baseline | 103.9 (32.05)
  Week 2 change from baseline: number analyzed (Participants) | 46
  Week 2 change from baseline | 3390.4 (1349.87)
  Week 4 change from baseline: number analyzed (Participants) | 44
  Week 4 change from baseline | 5308.9 (2073.59)
  Week 6 change from baseline: number analyzed (Participants) | 46
  Week 6 change from baseline | 6908.7 (3278.23)
  Week 8 change from baseline: number analyzed (Participants) | 44
  Week 8 change from baseline | 7319.3 (3587.14)
  Week 10 change from baseline: number analyzed (Participants) | 44
  Week 10 change from baseline | 7175.7 (4095.36)
  Week 12 change from baseline: number analyzed (Participants) | 42
  Week 12 change from baseline | 6446.3 (4422.46)
  Week 14 change from baseline: number analyzed (Participants) | 43
  Week 14 change from baseline | 6539.1 (4836.21)
  Week 16 change from baseline: number analyzed (Participants) | 42
  Week 16 change from baseline | 5316.6 (4941.13)
  Week 20 change from baseline: number analyzed (Participants) | 38
  Week 20 change from baseline | 3903.3 (4092.26)
  Week 24 change from baseline: number analyzed (Participants) | 36
  Week 24 change from baseline | 3190.2 (3172.22)
  Week 26 change from baseline: number analyzed (Participants) | 40
  Week 26 change from baseline | 3084.3 (2964.75)

ADVERSE EVENTS:
Time Frame: Day 1 up to final onsite visit (Week 26)
Description: The same event may appear as both a non-serious adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-06480605 500 mg IV
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 20/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06480605 500 mg IV (N=50)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2)
Peritonitis (Infections and infestations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06480605 500 mg IV (N=50)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Colitis ulcerative (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (7)
Nasopharyngitis (Infections and infestations) | 3 (3)
Pharyngitis (Infections and infestations) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT02840721/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT02840721/SAP_001.pdf